CLINICAL TRIAL: NCT06622252
Title: Intervention Development and Evaluation to Reduce Disparities in Quality of Life for Latino Families Impacted by Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Michelle Fortier, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20216922; ALS-5577146 (Other Grant/Funding Number: Alex's Lemonade Stand)
Record Dates: First submitted 2024-09-03; First posted 2024-10-02 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-02

CONDITIONS: Quality of Life; Pediatric Cancer; Caregiver Burden
MeSH Terms: conditions — Neoplasms; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: The first phase of this study involved qualitative and quantitative data collection and intervention feasibility testing using a single-arm within-subjects design.
  Our Community Based Participatory Research (CBPR) work to date has identified several barriers and targets for intervention.
  Accordingly, the newly designed intervention was split into three major components - Healthy Literacy, Caregiver Wellness, and Complementary Alternative Medicine. The second phase of this study is a preliminary randomized control trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Session (Corazones) Group (Experimental): Caregivers in this group will be asked to participate in a 13-session program (Corazones) delivered via Zoom. Caregivers will be asked to complete study questionnaires at the beginning of the study (Baseline), after completing the 13 zoom-based sessions (T2) and 3 months after participating in the program (T3). Caregivers will also be asked to participate in an interview with members of the research team to discuss their experiences participating in the program.
  Interventions: Other: 13-week session program
- Control Group (standard of care) (No Intervention): Caregivers will be asked to complete study questionnaires at the beginning of the study (Baseline), following week 2 of the intervention timeline, after week 12 of the intervention timeline (T2), and 3 months after the intervention groups completes their sessions (T3). Caregivers in this group will be offered the opportunity to participate in sessions after T3 surveys are completed. Attendance will not be compensated.

INTERVENTIONS:
Other: 13-week session program — The newly designed intervention was split into three major components - Healthy Literacy, Caregiver Wellness, and Culturally Competent Care and is delivered throughout a 13-session program delivered via Zoom. Sessions are guided by a psychologist, nutritionist, spirituality specialist, social worker, case coordinator, oncologist and traditional Chinese medicine practitioner. Sessions are intended for caregivers specifically, however, other members of the family may join if they choose to.
  Arms: Intervention Session (Corazones) Group

SUMMARY:
The purpose of this study is to determine if a culturally relevant caregiver intervention is effective in decreasing stress and improving quality of life in Spanish speaking Latino caregivers of children diagnosed with cancer compared to a control group.

DETAILED DESCRIPTION:
Phase 1:

Following informed consent, participants will be asked to complete measures at baseline, post intervention(T2), and 3 months post intervention (T3). Once baseline questionnaires are completed, subjects will participate in a 13-week intervention, comprised of live sessions aimed to address the components of, health literacy, caregiver wellness, and culturally competent care. Content of the sessions include culinary medicine, psycho-education, complementary alternative medicine, gardening, dance-based movement, question-answer forums and spirituality.

Participants will have access to a study specific a site which host recordings of all intervention sessions delivered throughout the intervention period and will track frequency and duration of video usage. Additionally, participants will have the opportunity to connect with each other outside of weekly sessions, using the chat feature within the video hosting platform.

All parts of the 13-session intervention will be delivered virtually via Zoom to ensure accessibility. Sessions will be scheduled on the dates and times most convenient for participants to encourage regular caregiver attendance. Zoom links will be shared with participants on a weekly basis via text or email. All sessions will be delivered in Spanish by native Spanish speakers with the exception of week 7 of the intervention. A translator will be present to facilitate this session.

Sessions are intended for caregivers specifically, however, other members of the family may join if they choose to. Sessions may require supplies for participant participation and engagement. In these circumstances the research team will provide supply kits to each participant. Additionally, participants will be loaned tablets as well as mobile hotspots throughout the intervention period to ensure equal opportunity for participation in this virtual pilot intervention. A member of the research team will be present at each session taking notes and assisting with any technical issue that may arise.

Immediately following the program, caregivers will be asked to participate in focus group or individual interview (qualitative) and to complete a measure of content and usability (quantitative) In addition the investigators will also interview our session experts/presenters to get their overall impressions of their intervention component. These interviews will be audio recorded.

Phase 2:

Procedures for phase 2 will remain the same for participants randomized to the intervention group. However, participants in the control group will only be asked to complete study questionnaires. To allow equal opportunity to control participants, caregivers will have the opportunity to attend intervention sessions after the 3 month follow up surveys are completed. Caregivers will not be compensated for attendance and sessions will not be recorded at this point.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of a Children's Hospital of Orange County (CHOC) oncology patient between the ages of 2-17 years old
* Caregiver of a CHOC oncology patient within 12 months of cancer diagnosis
* Caregiver of CHOC oncology patient must be able to speak and/or read and write in Spanish.
* Caregiver identifies as Latino

Exclusion Criteria:

* Presence of developmental disabilities, cognitive impairment, or severe psychiatric illness that would preclude participation in intervention sessions or interviews among caregivers and patients
* Caregiver unable to speak, read, and write in Spanish

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Parental Perceived Stress | baseline, immediately after the intervention, and 3 months post intervention
  Parental stress will be assessed using the Perceived Stress Scale (PSS). The PSS is a widely used 14-item self-report measure of perceived stress. Parents will be asked to rate statements such as "In the past month, how often have you been upset because of something that happened unexpectedly?" and "In the past month how often have you felt that things were going your way?" Subjects rate the items on a 5-point Likert-type scale with higher scores reflecting greater perceived stress. Seven items are reverse-keyed and items are summed to obtain the final score. Scores range from 0 -56 with higher scores indicating higher level of perceived stress. The PSS has been shown to have adequate reliability and validity
Parental emotional functioning (ANXIETY) | baseline, immediately after the intervention, and 3 months post intervention
  Parental emotional functioning will be measured using the Patient-Reported Outcome Measures (PROMIS) short form 8a (Anxiety). This form assesses 8 items of emotional stress and produces a standardized score ranging from 8-40 with higher raw scores signifying poorer emotional functioning.
Parental emotional functioning (DEPRESSION) | baseline, immediately after the intervention, and 3 months post intervention
  Parental emotional functioning will be measured using the Patient-Reported Outcome Measures (PROMIS) short form 8a (Depression). This form assesses 8 items of emotional stress and produces a standardized score ranging from 8-40 with higher raw scores signifying poorer emotional functioning.
Parental Quality of Life | baseline, immediately after the intervention, and 3 months post intervention
  Parental quality of life (Health Survey) will be assessed using the Medical Outcomes Survey (MOS Short Form-36), which is a widely used measure of both physical and mental functioning. scores range from 0-100 with lower scores representing more disability. The higher the score the less disability. Reliability and validity are good.

CONTACTS AND LOCATIONS:
Locations (1):
- CHOC Children's, Orange, California, United States